CLINICAL TRIAL: NCT06732427
Title: Efficacy and Safety of Fospropofol Disodium for Injection in the Painless Endoscopic Diagnosis and Treatment: a Multicenter-prospective, Randomized, Controlled Trial
Brief Title: Clinical Study of Fospropofol Disodium for Injection in the Painless Endoscopic Diagnosis and Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Collaborators: Rugao People's Hospital (Other); Qidong People's Hospital (Unknown); Hai 'an People's Hospital (Unknown); Rudong County Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-YCRF-M1021
Record Dates: First submitted 2024-12-06; First posted 2024-12-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-11

CONDITIONS: Efficacy and Safety
Keywords: Painless gastrointestinal endoscopy; fospropofol disodium for injection
MeSH Terms: interventions — fospropofol; Injections; Sufentanil; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Using a computer-generated randomized number table, the patients were divided into two groups: group L (fospropofol disodium group) and group B (propofol group). After determining the group of enrolled patients, the drug was administered by two fixed anesthesiologists. The study drug is prepared by someone who do not participate in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fospropofol Disodium (Experimental): Painless gastrointestinal endoscopy in group L was mainly performed using fospropofol Disodium for injection
  Interventions: Drug: fospropofol Disodium for injection
- propofol (Active Comparator): Painless gastrointestinal endoscopy in group B was mainly performed using propofol
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: fospropofol Disodium for injection — Group L received slow intravenous sufentanyl 0. 1 ug / kg +fospropofol Disodium for injection 8mg / kg (completed within 60 seconds)
  Other Names: sulfentanyl
  Arms: Fospropofol Disodium
Drug: Propofol — Group B received slow intravenous sufentanyl 0. 1 ug / kg +propofol 2mg / kg (completed within 60 seconds)
  Other Names: sulfentanyl
  Arms: propofol

SUMMARY:
This is a study on the efficacy and safety of fospropofol disodium for injection in painless endoscopic diagnosis and treatment, project No.2024-YCRF-M1021, which will take more than 2 years to complete.

This is a multicenter, randomized, double-blind, controlled clinical study. Using a computer-generated randomized number table, the patients were divided into two groups: the group L (fospropofol disodium group) and the group B (propofol group). After determining the group of enrolled patients, the drug was administered by two fixed anesthesiologists By participating in this study, it is possible to make your anesthesia induction stable, stable intraoperative circulation, awake and safe and comfortable, to reduce the incidence of intraoperative hypoxemia, intraoperative awareness, cardiovascular and cerebrovascular malignant events (malignant arrhythmia, cardiac arrest), which is conducive to your rapid postoperative recovery and reduce hospitalization costs.

DETAILED DESCRIPTION:
1. Research background: Painless endoscopic diagnosis and treatment technology refers to letting patients undergo various examinations and treatments in a comfortable and painless state, including painless gastrointestinal endoscopy, painless abortion, painless hysteroscopy, etc. These diagnosis and treatment operations are widely carried out in the outpatient department. The development of painless diagnosis and treatment technology has greatly improved the patient's satisfaction and comfort level. Anesthesia is the leading discipline of painless diagnosis and treatment technology. In recent years, the development of painless technology of intravenous general anesthesia and the selection of general anesthesia drugs have been controversial areas. It is very important to determine an appropriate anesthesia scheme.

   It has been reported that the incidence of propofol in the diagnosis and treatment of painless gastroscopy reached 8.4%. For adult patients sedated by propofol, the dosage of propofol gradually decreased with the age of patients, and the incidence of hypoxemia increased, accompanied by the overall trend of increasing adverse cardiovascular events. To achieve rapid and predictable recovery requires stable intraoperative respiratory circulation, stable recovery, and reduced adverse reactions such as postoperative nausea, vomiting and injection pain, while propofol is easy to cause injection pain at the injection site of patients.

   Fospropofol disodium for injection is an effective intravenous sedative hypnotic agent that was approved by the United States Food and Drug Administration (FDA) in December 2008 for adult anesthesia monitoring undergoing diagnosis or treatment process. It gradually releases the active metabolite propofol, with slow onset and more stable breathing and circulation. In 2021, the fospropofol disodium for injection copied by Yichang Renfu Pharmaceutical Co. Ltd. was approved by the human bioequivalence study (BE). The fospropofol disodium for injection developed by Chinese scholars is different from American scholars, with better drug structure and better drug specifications. Fospropofol disodium for injection is a chemical class 1 new drug, which is one of the most advanced systemic intravenous anesthetics studied at home and abroad.

   In the Guidance on clinical Application of fospropofol disodium for injection published by the Chinese Journal of Anesthesiology, the indication has been approved as the induction of general anesthesia in adults. Phase Ⅲ clinical trials suggest that the efficacy of Fospropofol disodium for injection is more stable in the process of anesthesia induction to maintenance, and its efficacy duration is long, which can save the amount of subsequent sedative and analgesic drugs, meet the actual clinical needs and meet the requirements of pharmacoeconomics. In the pre-experiment, our research group found that 7.5 -8.5mg / kg fospropofol disodium for injection was used for anesthesia with painless gastrointestinal endoscopy, with definite effect, slight respiratory depression and stable hemodynamics.
2. The purpose of this study: Observe the safety and effectiveness of fospropofol disodium for injection in painless gastrointestinal endoscopic diagnosis and treatment, optimize the clinical anesthesia scheme, and provide reference for clinical medication for comfortable diagnosis and treatment.
3. Research method: This is a multicenter, randomized, double-blind, controlled clinical study. Using a computer-generated randomized number table, the patients were divided into two groups: the group L (fospropofol disodium group) and the group B (propofol group). After determining the group of enrolled patients, the drug was administered by two fixed anesthesiologists. Mainly observe the success rate of sedation, total amount of fospropofol disodium for injection and propofol, additional doses, the occurrence of intraoperative hypoxemia, intraoperative circulatory system such as hypotension, hypertension, bradycardia, tachycardia, intraoperative adverse reactions such as reflex cough, intraoperative body movement, injection pain, postoperative recovery quality and other adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-65 years, weight 40-65kg, male or female;
2. Patients undergoing painless gastrointestinal endoscopy or painless colonoscopy;
3. American Society of Anesthesia (ASA) grades I-II;
4. Patients and their families can understand and fill in various rating scales, and voluntarily sign the informed consent form; -

Exclusion Criteria:

1. Patients with simple and painless gastroscopy
2. Allergy to this study drug and any ingredients;
3. Patients with pathological obesity / obstructive sleep apnea, patients with difficult respiratory tract management;
4. Acute upper respiratory tract infection and asthma attacks;
5. Liver and kidney insufficiency, abnormal heart function;
6. History of mental disorders, long-term use of analgesics; history of drug addiction and drug use;
7. Do not voluntarily cooperate with the patient or be unsuitable by the investigator to participate in the trial.-

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sedation success rate | At 5 minutes after anesthetic administration
  Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score ≤ 1(The rating scale ranges from levels 0 to 5, and lower MOAA / S score indicates deeper depth of sedation, namely a higher scores mean a worse outcome.) or EEG bispectral index (BIS) value <64( The rating scale ranges from levels 0 to 100, and lower BIS score indicates deeper depth of sedation, namely a higher scores mean a worse outcome. )within 5 minutes (no additional drug within 5 minutes)
Length of successful induction of anesthesia | During anesthesia
  Time from the first start of administration of study drug to Modified Observer's Assessment of Alertness/Sedation score ≤1 ((The rating scale ranges from levels 0 to 5, and lower MOAA / S score indicates deeper depth of sedation, namely a higher scores mean a worse outcome.) or EEG bispectral index (BIS) value <64(The rating scale ranges from levels 0 to 100, and lower BIS score indicates deeper depth of sedation, namely a higher scores mean a worse outcome. )
hypoxaemia | During anesthesia
  Oxygen saturation below 90% over 30 seconds or requires any type of airway assistance (including jaw support, artificial airway)

SECONDARY OUTCOMES:
Hemodynamic index | During anesthesia
  The occurrence of hypotension, hypertension, bradycardia, and tachycardia
Limb movements of the patient during the operation | During anesthesia
  No movement of limbs (10 points); slight movement, occasionally (8 points); slight movement, frequent (6 points), vigorous movement, arms and legs only (4 points); vigorous body and head movement (2 points)
Wake up time | During anesthesia
  Time from the end of surgery until Modified Observer's Assessment of Alertness/Sedation score=5 points(The rating scale ranges from levels 0 to 5, and lower MOAA / S score indicates deeper depth of sedation, namely a higher scores mean a worse outcome).
Awakening quality of anesthesia | 10 minutes ,20 minutes and 30 minutes after awakening
  Wake quality was assessed using a modified AIdrete score(The rating scale ranges from levels 0 to 10, and the lower the score indicates that the worse the recovery mass, namely a higher scores mean a better outcome).
Total amount of study drug used | During anesthesia
  Total dosage of fospropofol disodium and propofol for injection, and number of additional doses

OTHER OUTCOMES:
General data of the patient(1) | Preoperative and intraoperative
  age
General data of the patient(2) | Preoperative and intraoperative
  height
General data of the patient(3) | Preoperative and intraoperative
  weight
General data of the patient(4) | Preoperative and intraoperative
  Other general data, including gender, current medical history, history of combined diseases and medication allergy, history of hypertension / diabetes (most hypertension / blood glucose, type and age of medication, and presence of other organs); mouth opening, the history of snoring, history of Obstructive sleep apnea and hypopnea syndrome, number of shots of gastrointestinal endoscopy, basic blood oxygen value
Perioperative adverse effects | up to 24 hours after surgery
  Including intraoperative awareness, injection pain, nausea, vomiting, itching, and paraesthesia
Evaluation of patient satisfaction with anesthesia | up to 24 hours after surgery
  The rating scale ranges from levels dissatisfaction, basic satisfaction, satisfaction to very satisfaction, the higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao MB Director of scientific research Department, Doctor, Principal Investigator — The Affiliated Hospital of Nantong University
Locations (5):
- China (5):
  - Hai 'an People's Hospital, Hai’an, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Qidong People's Hospital, Qidong, Jiangsu
  - Rudong County Hospital of Traditional Chinese Medicine, Rudong, Jiangsu
  - Rugao People's Hospital, Rugao, Jiangsu

IPD SHARING:
Plan to Share IPD: No